CLINICAL TRIAL: NCT06258577
Title: Screening for Gaucher Disease and Acid Sphingomyelinase Deficiency From Taiwanese Candidates With Splenomegaly and/or Thrombocytopenia
Brief Title: Screening for Gaucher Disease and Acid Sphingomyelinase Deficiency
Status: Not yet recruiting | Type: Observational
Sponsor: Chung-Hsing Wang (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Chung-Hsing Wang, Attending Physicians, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Other Study IDs: CMUH112-REC2-098
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- candidates: In the first phase, patients with hepatosplenomegaly of unknown etiology will be initially screened using an electronic medical record database, and in the second phase, laboratory analysis of biomarkers, including Dry blood spot (DBS) for GBA1 enzyme activity, plasma Lyso-GB1 levels and GBA1 gene sequencing, will be performed.
- control: Compare the blood test with the candidates group.

SUMMARY:
High-risk screening for Gaucher disease and Acid Sphingomyelinase Deficiency in patients with splenomegaly and/or thrombocytopenia in Taiwan

DETAILED DESCRIPTION:
Late-onset Gaucher disease (GD) present a unique set of challenges compared to their early-onset counterparts. Symptoms may not appear until adulthood, leading to delayed diagnosis and treatment. This delay can result in irreversible damage to affected tissues and organs, such as the liver, spleen, and central nervous system. Additionally, many late-onset GD are underdiagnosed or misdiagnosed due to their rarity and the variability of symptoms. This study is divided into two phases. In the first phase, patients with hepatosplenomegaly of unknown etiology will be initially screened using an electronic medical record database, and in the second phase, laboratory analysis of biomarkers, including Dry blood spot (DBS) for GBA1 enzyme activity, plasma Lyso-GB1 levels and GBA1 gene sequencing, will be performed. Acid sphingomyelinase deficiency (ASMD) is another lysosomal storage disorder that shares symptoms with GD. Consistent with the above screening strategy for GD patients in two phases (DBS for ASM enzyme activity, plasma Lyso-SM levels and ASM gene sequencing). This study will involve 2,000 candidates from electronic healthcare databases, 240 patients from outpatient clinics, and a cohort of 6 GD1/GD3 patients as controls. In conclusion, initial screening for late-onset GD and ASMD can provide patients with treatment opportunities that can improve outcomes for those affected by these rare diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of splenomegaly
2. Clinical diagnosis of thrombocytopenia

Exclusion Criteria:

1. Clinical diagnosis of gaucher disease
2. Clinical diagnosis of acid sphingomyelinase
3. Clinical diagnosis of malignant tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient of gaucher disease or acid sphingomyelinase
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Confirmation of Disease | 1 month
  DBS for GBA1 enzyme activity or ASM enzyme activity positive、GBA1 gene sequencing or ASM gene sequencing positive

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Hsing Wang, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospita, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wan L, Hsu CM, Tsai CH, Lee CC, Hwu WL, Tsai FJ. Mutation analysis of Gaucher disease patients in Taiwan: high prevalence of the RecNciI and L444P mutations. Blood Cells Mol Dis. 2006 May-Jun;36(3):422-5. doi: 10.1016/j.bcmd.2006.02.001. Epub 2006 Mar 20. PMID 16546416
- [Result] Revel-Vilk S, Fuller M, Zimran A. Value of Glucosylsphingosine (Lyso-Gb1) as a Biomarker in Gaucher Disease: A Systematic Literature Review. Int J Mol Sci. 2020 Sep 28;21(19):7159. doi: 10.3390/ijms21197159. PMID 32998334
- [Result] Pinto C, Sousa D, Ghilas V, Dardis A, Scarpa M, Macedo MF. Acid Sphingomyelinase Deficiency: A Clinical and Immunological Perspective. Int J Mol Sci. 2021 Nov 28;22(23):12870. doi: 10.3390/ijms222312870. PMID 34884674
- [Result] McGovern MM, Avetisyan R, Sanson BJ, Lidove O. Disease manifestations and burden of illness in patients with acid sphingomyelinase deficiency (ASMD). Orphanet J Rare Dis. 2017 Feb 23;12(1):41. doi: 10.1186/s13023-017-0572-x. PMID 28228103
- [Result] Jones SA, McGovern M, Lidove O, Giugliani R, Mistry PK, Dionisi-Vici C, Munoz-Rojas MV, Nalysnyk L, Schecter AD, Wasserstein M. Clinical relevance of endpoints in clinical trials for acid sphingomyelinase deficiency enzyme replacement therapy. Mol Genet Metab. 2020 Sep-Oct;131(1-2):116-123. doi: 10.1016/j.ymgme.2020.06.008. Epub 2020 Jun 24. PMID 32616389
- [Result] Loftus WK, Metreweli C. Normal splenic size in a Chinese population. J Ultrasound Med. 1997 May;16(5):345-7. PMID 9315173